CLINICAL TRIAL: NCT03307603
Title: A Phase Ib/II Study of Yttrium-90 Radioembolization With Nivolumab for Treatment of Liver and Extra-hepatic Metastases From Colorectal Cancer
Brief Title: Yttrium-90 Radioembolization + Nivolumab for Liver + Extra-hepatic Metastases From Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor chose not to continue
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3216
Record Dates: First submitted 2017-09-07; First posted 2017-10-11 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Yttrium-90 radioembolization; Nivolumab
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Yttrium-90 + Nivolumab (Experimental): 240 mg Nivolumab intravenously, beginning at 2 weeks after Yttrium-90 treatment and given every 2 weeks until progression or toxicity. Additional dose at 2 weeks prior to Y-90 will be given if the first 3 patients do not have toxicity. If any of the first 3 patients have toxicity, the schedule can be relaxed to begin 3 weeks after Y-90 treatment.
  Interventions: Radiation: yttrium-90 radioembolization; Drug: Phase Ib - nivolumab; Drug: Phase II - nivolumab

INTERVENTIONS:
Radiation: yttrium-90 radioembolization — Yttrium-90 will be given as biocompatible resin-based microspheres and will be introduced to the tumor(s) on one side of the liver through a catheter placed in the right or left hepatic artery. The dose of radiation will be determined by a radiologist and will be based on body surface area and tumor burden.
Drug: Phase Ib - nivolumab — 240 mg intravenously
Drug: Phase II - nivolumab — nivolumab will be administered as determined during the phase Ib portion of the study. Nivolumab will be administered on an every 2 week basis for a total of 48 weeks or until disease progression, unacceptable toxicity or discontinuation due to patient/physician preference.

SUMMARY:
This study has two portions. The main goal of the Phase Ib portion of this research study is to see at what time Yttrium-90 (Y-90) radioembolization therapy and nivolumab can safely be given to patients without having too many side effects. Other purposes of this research study will be to study any tumor responses.

The Phase II portion of the study will test how many patients show shrinkage in their tumor with this combination of medicines and what changes occur inside the cancer cells and blood cells after treatment. The study team will pick the part of the study each subject participates in.

Y-90 radioembolization therapy is minimally invasive procedure that combines two types of therapy (embolization which blocks certain blood vessels, and radiation therapy, which kills cancer cells) to treat cancer tumors in the liver. This works with tiny glass or resin beads filled with the radioactive isotope yttrium-90 (Y-90). They are placed inside the blood vessels that feed the tumor in the liver. This blocks the supply of blood to the cancer cells and delivers a high dose of radiation to the tumor while sparing normal tissue.

Nivolumab is an FDA approved medicine that is used for the treatment of different types of cancers and metastases (second growths from cancer).

DETAILED DESCRIPTION:
Primary Objective

Phase Ib: To determine the safety and tolerability of Y-90 radioembolization therapy when given in conjunction with neoadjuvant/adjuvant nivolumab as assessed by CTCAE version 4, in patients with metastatic colorectal cancer who undergo Y-90 radioembolization to hepatic metastases and have additional disease located outside of the radioembolization field.

Phase II: To determine the objective response rate (RR) as assessed by RECIST criteria of metastases located outside of the Y-90 radioembolization treatment field in patients with metastatic colorectal cancer who undergo Y-90 radioembolization to hepatic metastases and receive neoadjuvant/adjuvant nivolumab.

Secondary Objectives

Phase Ib:

To assess the response rate (RR) of patients with metastatic colorectal cancer who undergo standard Y-90 radioembolization therapy to hepatic metastases as well as neoadjuvant/adjuvant nivolumab as assessed by measurement of foci located outside of the Y-90 radioembolization field.

Phase II:

To assess the progression free survival (PFS) of patients with metastatic colorectal cancer who undergo standard Y-90 radioembolization therapy to hepatic metastases as well as neoadjuvant/adjuvant nivolumab as assessed by measurement of metastatic foci located outside of the Y-90 radioembolization field.

To assess the 1-year and 2-year overall survival (OS) rate of patients with metastatic colorectal cancer who undergo standard Y-90 radioembolization therapy to hepatic metastases as well as neoadjuvant/adjuvant nivolumab.

Correlative Objectives

To characterize the baseline expression and localization of immune markers including Programmed cell death protein 1 (PD-1), Programmed cell death protein ligand 1 (PD-L1), Programmed cell death protein ligand 2 (PD-L2), T-cell immunoglobulin and mucin-domain containing-3 (TIM-3), Lymphocyte activation gene 3 (LAG-3), Tumor necrosis factor receptor superfamily, member 4 (OX40) and Cluster of Differentiation 137 (CD137) within the tumor microenvironment and correlate this with treatment response.

To examine the change in density of Cluster of Differentiation (CD8)+/Kiel-67 (Ki-67) high tumor infiltrating lymphocytes and expression levels of PD-L1 in the tumor parenchyma prior to and following treatment with Y-90 and nivolumab as assessed in a lesion outside of the radioembolization field. Changes in biomarkers will be correlated with treatment response.

To assess baseline and changes in the immune signature of Y-90 naïve colorectal cancer in patients with liver metastases who receive Y-90 radioembolization and nivolumab therapy. Human transcriptome gene expression arrays will be performed and expression data will be used to identify immune cell subsets using CIBERSORT and immune signatures will be assessed using ImmuneSigDB.

To assess baseline and changes in non-targeted tumor antigens using Proto Array Human Protein MicroArray Profiling and Immunoglobulin G (IgG) quantification in patients with liver metastases who receive Y-90 radioembolization and nivolumab therapy. Changes in profile will be correlated with treatment response.

Study Design

This is a single arm phase Ib/II trial assessing the safety and toxicity (phase Ib) followed by the antitumor activity (response rate) (phase II) of nivolumab when administered in combination with Y-90 radioembolization therapy.

Study design

Eligible patients will undergo Y-90 radioembolization to one side of the liver according to standard practice as directed by an interventional radiologist. Yttrium-90 will be given as biocompatible resin-based microspheres and will be introduced to the tumor(s) on one side of the liver through a catheter placed in the right or left hepatic artery (depending on the lobe treated). The dose of radiation will be determined by a radiologist and will be based on body surface area and tumor burden. During the phase Ib portion of the study, nivolumab will be administered per the scheduling algorithm at a flat dose of 240 mg intravenously over 30 +/- 5 minutes. Depending on the schedule being assessed, this may include a neoadjuvant dose to be given prior to Y-90, and will contain an adjuvant dose following Y-90 therapy. During the phase II portion of the study, nivolumab will be administered as determined during the phase Ib portion of the study. Nivolumab will continue to be administered on an every 2 week basis for a total of 48 weeks or until disease progression, unacceptable toxicity or discontinuation due to patient/physician preference. Patients will be evaluated with a history and physical exam as well as laboratory parameters once every 2 weeks throughout the duration of the study. Patients will undergo CT scans of the chest and pelvis as well as MRI of the liver to assess disease status 2 months following the Y-90 radioembolization procedure, then every 3 months for a total of 2 years. Upon completing treatment, patients will be followed monthly for another 100 days for toxicity monitoring. Archived tissue specimens will be obtained at baseline and a post-treatment biopsy of a metastatic lesion located outside of the Y-90 radioembolization field will be obtained 60 +/- 5 days following treatment with Y-90 radioembolization for assessment of intratumoral immunogenicity. Carcinoembryonic antigen (CEA) levels will be assessed at baseline, then once monthly for 6 months, then every 3 months for a total of 2 years. Patients will have a pre-treatment serum sample collected as well as post-treatment samples collected approximately 6 weeks, 12 weeks and 20 weeks after treatment with Y-90 radioembolization for banking, to be used in the future assessment of putative biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic colorectal cancer.
* Patients must have liver metastases and be appropriate for treatment with Y-90 radioembolization therapy as determined by the treating medical oncologist and interventional radiologist. Prior Y-90 therapy is not permitted.
* Patients must have measurable disease that is located outside of the Y-90 radioembolization field.
* Patients must have a metastatic focus amenable to biopsy that is located outside of the Y-90 radioembolization field. It is permissible to use the same lesion for biopsy as for assessment to tumor response.
* Patients must have received at least one line of prior chemotherapy and must have had resolution of all side effects to at least at Grade 1 prior to trial entry.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Patients must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dl
  * Leukocytes ≥ 2,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except in patients with Gilbert Syndrome, who can have a total bilirubin < 3.0 mg/dL)
  * Aspartate aminotransferase (AST) (SGOT) ≤ 3 X institutional upper limit of normal
  * Alanine aminotransferase (ALT) (SGPT) ≤ 3 X institutional upper limit of normal
  * Serum creatinine ≤ 1.5 X ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 1.00/ 72 x serum creatinine in mg/dL

Male CrCl = (140 - age in years) x weight in kg x 1.00/ 72 x serum creatinine in mg/dL

-Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. Women of childbearing potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mili-international units/milliliter (mIU/mL).

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, with have a failure rate of < 1% when used consistently and correctly.

* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception).
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with ongoing toxicities > grade 1 according to NCI CTCAE Version 4.0 (excluding alopecia and neuropathy) due to prior anti-cancer therapy.
* Patients receiving any other investigational agent or active chemotherapy.
* Patients who have previously been treated an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-Cytotoxic T-lymphocyte associated protein (CTLA)-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Patients with a known autoimmune disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Patients having a condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg/day prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients who are positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection.
* Patients with a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Patients who have received prior external beam radiation therapy to the liver.
* Patients who have clinical evidence of ascites or are in clinical liver failure.
* Patients who are known to have greater than 20% lung shunting of the hepatic artery blood flow determined by Technetium microaggregated albumin (MAA) scan (if conducted prior to study enrollment).
* Patients who have had a standard of care pre-assessment angiogram that demonstrates abnormal vascular anatomy that would result in significant reflux of hepatic arterial blood to the stomach, pancreas or bowel.
* Patients with known portal vein thrombosis.
* Patients with untreated brain metastases or leptomeningeal metastases will be excluded. Patients with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are pregnant or breastfeeding will be excluded from the study due to the potential teratogenic or abortifacient effects that may result from nivolumab or Y-90 Theraspheres. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab and Y-90, breastfeeding should be discontinued if the mother is treated with nivolumab and Y-90. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with nivolumab. In addition, these subjects are at increased risk of lethal infections when treated with immunosuppressive agents. Screening HIV testing is not required.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Phase I: Average number of serious adverse events experience by patients | Up to 2 years after starting study
  assessed by CTCAE version 4 of nivolumab in combination with Y-90 radioembolization when administered to patients with metastatic colorectal cancer who have hepatic metastases appropriate for treatment with Y-90 radioembolization therapy.
Phase II: Response rate | Up to 2 years after starting study
  assessed by RECIST 1.1 criteria of metastases outside of the Y-90 radioembolization treatment field in patients with metastatic colorectal cancer who undergo Y-90 radioembolization therapy to hepatic metastases followed by nivolumab.

SECONDARY OUTCOMES:
Phase I: Progression free survival (PFS) | Up to 2 years after starting study
  Progression free survival (PFS) of patients with metastatic colorectal cancer who undergo standard Y-90 radioembolization therapy to hepatic metastases followed by nivolumab as assessed by metastatic foci located outside of the Y-90 radioembolization field.
Phase I: Overall survival | Up to 2 years after starting study
  Overall survival of patients with metastatic colorectal cancer who undergo standard Y-90 radioembolization therapy to hepatic metastases followed by nivolumab.
Phase II: Progression free survival (PFS) | Up to 2 years after starting study
  Progression free survival (PFS) of patients with metastatic colorectal cancer who undergo standard Y-90 radioembolization therapy to hepatic metastases followed by nivolumab as assessed by metastatic foci located outside of the Y-90 radioembolization field.
Phase II: Overall survival | Up to 2 years after starting study
  Overall survival of patients with metastatic colorectal cancer who undergo standard Y-90 radioembolization therapy to hepatic metastases followed by nivolumab.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Eads, MD, Principal Investigator — University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center